CLINICAL TRIAL: NCT03092531
Title: Adaptive Intervention Strategies Trial for Strengthening Adherence to Antiretroviral HIV Treatment Among Youth
Brief Title: Positive Steps to Enhance Problem Solving Skills
Acronym: STEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Matthew Mimiaga, ScD, MPH, MA, Professor of Epidemiology, UCLA Fielding School of Public Health, and Psychiatry & Biobehavioral Sciences, UCLA David Geffen School of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01NR017098-01A1 (NIH)
Record Dates: First submitted 2017-03-10; First posted 2017-03-28 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Adherence
Keywords: HIV; ART Adherence; Adolescents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Block randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive STEPS (Experimental): Step 1) all participants randomized to the experimental condition will receive low-intensity, daily two-way SMS texts of personalized reminders to take medications as prescribed ("social-cognitive cues"). If a participants demonstrates >90% adherence they will remain on step one. Participants who continue to have difficulty adhering to their HIV medications at one month after baseline or anytime up to the end of month three (weeks five through twelve) will progress to Step 2) Five in-person, counseling sessions. Each counseling session will last approximately 50 minutes.
  Interventions: Behavioral: Positive STEPS
- Standard of Care (No Intervention): The standard health services offered at each site (e.g., mental health services, case management) and a brief adherence educational session. This will consist of a review of medications and recommended dosing (i.e., to understand regimen), adherence expectations, toxicity expectations and medication misperceptions.The participant will then view a 20-minute animated tutorial which explains the importance of adherence to antiretroviral medication effectiveness.

INTERVENTIONS:
Behavioral: Positive STEPS — Step 1: 2 way SMS text messages; Step 2: Five in-person, counseling sessions. Each counseling session will last approximately 50 minutes.
  Arms: Positive STEPS

SUMMARY:
This randomized control trial is to test the efficacy of a stepped-care "adaptive" Antiretroviral Therapy (ART) adherence intervention ("Positive STEPS") for HIV infected adolescents and young adults, ages 16 to 29. Stepped care is a healthcare delivery model in which the least resource intensive part of an intervention is delivered first, and only those who do not improve then receive the high intensity, more resource intensive part of an intervention.

DETAILED DESCRIPTION:
HIV infected adolescents and young adults will be recruited from Providence, Rhode Island, Boston, Massachusetts and Chicago, Illinois. Participants will be equally randomized to:

1. "Positive STEPS" - a stepped care, adherence intervention with integrated technology (2-way daily text messaging aimed at improving ART adherence). If text messaging is not sufficient to overcome the barriers to ART adherence;these individuals will then also receive the more intensive component based on general principles of cognitive-behavioral therapy.
2. Standard of Care comparison group including a brief adherence educational session. This will consist of a review of medications and recommended dosing (i.e., to understand regimen), adherence expectations, toxicity expectations and medication misperceptions.The participant will then view a 20-minute animated tutorial which explains the importance of adherence to antiretroviral medication effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Between 16 and 29 years of age
* HIV-infected (perinatally, transfusion, or behaviorally-acquired)
* Currently taking or prescribed antiretroviral therapy and: 1) Began taking ART < 3 months ago, OR 2) Has been taking ART for >3 AND has missed one or more doses in the past week or more than 3 doses in the past month.
* Daily access to a cell phone
* Has lived in the greater Providence, Boston, or Chicago area greater than three months
* Self-reports < 90% ART medication adherence in the past month (i.e., missed one or more doses in the past week or more than 3 doses in the past month) at screening
* Able to speak and understand English
* Not currently enrolled in another ART-adherence intervention study
* Willing and able to complete all study visits in person or remotely via video conferencing platform

Exclusion Criteria:

* Unable to give informed consent due to severe mental or physical illness, cognitive limitation, or substance intoxication at baseline visit
* HIV-uninfected
* Not currently on antiretroviral therapy
* Does not own a cell phone
* Has lived in the greater Providence, Boston, or Chicago area for less than three months or is planning to move outside the area within the next year
* Self-reports > 90% ART medication adherence in the past month AND has been taking ART for more than 3 months
* Unable to speak and understand English
* Currently enrolled in another ART-adherence intervention study
* Not willing to and able to complete all study visits in person or remotely via video conferencing platform

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 123 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Reduced HIV Viral Load | Baseline, 4 month, 8 month, 12 month
  Blood specimen collection tested for HIV Viral Load
ART Medication Level in Hair Sample | Baseline, 4 month, 8 month, 12 month
  Collection of hair sample to measure level of ART
Daily ART adherence | 4 month, 8 month, 12 month
  Monitoring of Wisepill device for electronic adherence data
Daily ART Adherence | Baseline, 4 month, 8 month, 12 month
  Self report via research assessment

SECONDARY OUTCOMES:
Reduced HIV Symptoms | Baseline, 4 month, 8 month, 12 month
  Medical record review for increase or decrease in symptoms associated with HIV
Engagement in HIV Care | Baseline, 4 month, 8 month, 12 month
  Number of kept versus number of scheduled visits verified by medical record
Medication changes to ART | Baseline, 4 month, 8 month, 12 month
  Verified by medical record

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Mimiaga, ScD, MPH, Principal Investigator — UCLA, School of Public Health, Department of Epidemiology, Fielding School of Public Health; Robert Garofalo, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (4):
- United States (4):
  - UCLA Center for LGBTQ+ Advocacy, Research & Health, Los Angeles, California
  - Lurie Childrens Hospital, Chicago, Illinois
  - Fenway Health Institute, Boston, Massachusetts
  - Brown University School of Public Health, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Present at least annually on data collected after the second year when sufficient baseline data is collected. Randomized controlled efficacy trial, we anticipate that most of the papers and data-based projects and presentations will happen in year 5, once baseline data and follow-up assessments have occurred. Sharing findings will involve several papers, including a baseline paper, intervention-specific paper, primary paper describing the study outcomes, secondary outcomes papers and potentially a book that describes the intervention, submitting to lead workshops on the intervention approach at relevant national and international meetings and conferences. Raw data for additional analysis will be available by contacting the Principal Investigators.

REFERENCES:
- [Derived] Klasko-Foster LB, Biello KB, Lodge W 2nd, Olson J, Mimiaga MJ. Transitioning from Face to Face to the Digital Space: Best Practices and Lessons Learned Leveraging Technology to Conduct HIV-Focused Interventions. Telemed J E Health. 2022 Jul;28(7):1070-1073. doi: 10.1089/tmj.2021.0190. Epub 2022 Jan 6. PMID 34995162
- [Derived] Mimiaga MJ, Kuhns LM, Biello KB, Olson J, Hoehnle S, Santostefano CM, Hughto JMW, Safi H, Salhaney P, Chen D, Garofalo R. Positive STEPS - a randomized controlled efficacy trial of an adaptive intervention for strengthening adherence to antiretroviral HIV treatment among youth: study protocol. BMC Public Health. 2018 Jul 13;18(1):867. doi: 10.1186/s12889-018-5815-9. PMID 30001703

DOCUMENTS (1):
  • Informed Consent Form (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03092531/ICF_000.pdf